CLINICAL TRIAL: NCT06712316
Title: A Phase II/III, Multisite, Randomized Master Protocol for a Global Trial of BNT327 in Combination With Chemotherapy and Other Investigational Agents in First-line Non-small Cell Lung Cancer
Brief Title: Safety, Efficacy, and Pharmacokinetics of BNT327 in Combination With Chemotherapy and Other Investigational Agents for Lung Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BNT327-06; 2024-515764-31-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-11; First posted 2024-12-02 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: First-line treatment; Combination with chemotherapy; Combination with other investigational agents; Bispecific antibody; Programmed death-ligand 1 (PD-L1); Vascular endothelial growth factor (VEGF) A; Immunotherapy; Programmed Death-1 monoclonal antibodies
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Carboplatin; Pemetrexed; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Substudy A Phase 2 - Pumitamig Dose 1 + Carboplatin + Pemetrexed (Experimental)
  Interventions: Drug: Pumitamig; Drug: Carboplatin; Drug: Pemetrexed
- Substudy A Phase 2 - Pumitamig Dose 2 + Carboplatin + Pemetrexed (Experimental)
  Interventions: Drug: Pumitamig; Drug: Carboplatin; Drug: Pemetrexed
- Substudy A Phase 3 - Pumitamig + Carboplatin + Pemetrexed (Experimental): Pumitamig dose 3 for Phase 3
  Interventions: Drug: Pumitamig; Drug: Carboplatin; Drug: Pemetrexed
- Substudy A Phase 3 - Pembrolizumab + Carboplatin + Pemetrexed (Active Comparator)
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Pemetrexed
- Substudy B Phase 2 - Pumitamig Dose 1 + Carboplatin + Paclitaxel (Experimental)
  Interventions: Drug: Pumitamig; Drug: Carboplatin; Drug: Paclitaxel
- Substudy B Phase 2 - Pumitamig Dose 2 + Carboplatin + Paclitaxel (Experimental)
  Interventions: Drug: Pumitamig; Drug: Carboplatin; Drug: Paclitaxel
- Substudy B Phase 3 - Pumitamig + Carboplatin + Paclitaxel (Experimental): Pumitamig dose 3 for Phase 3
  Interventions: Drug: Pumitamig; Drug: Carboplatin; Drug: Paclitaxel
- Substudy B Phase 3 - Pembrolizumab + Carboplatin + Paclitaxel (Active Comparator)
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Pumitamig — Intravenous infusion
  Other Names: BNT327
  Arms: Substudy A Phase 2 - Pumitamig Dose 1 + Carboplatin + Pemetrexed; Substudy A Phase 2 - Pumitamig Dose 2 + Carboplatin + Pemetrexed; Substudy A Phase 3 - Pumitamig + Carboplatin + Pemetrexed; Substudy B Phase 2 - Pumitamig Dose 1 + Carboplatin + Paclitaxel; Substudy B Phase 2 - Pumitamig Dose 2 + Carboplatin + Paclitaxel; Substudy B Phase 3 - Pumitamig + Carboplatin + Paclitaxel
Drug: Pembrolizumab — Intravenous infusion
  Arms: Substudy A Phase 3 - Pembrolizumab + Carboplatin + Pemetrexed; Substudy B Phase 3 - Pembrolizumab + Carboplatin + Paclitaxel
Drug: Carboplatin — Intravenous infusion
Drug: Pemetrexed — Intravenous infusion
  Arms: Substudy A Phase 2 - Pumitamig Dose 1 + Carboplatin + Pemetrexed; Substudy A Phase 2 - Pumitamig Dose 2 + Carboplatin + Pemetrexed; Substudy A Phase 3 - Pembrolizumab + Carboplatin + Pemetrexed; Substudy A Phase 3 - Pumitamig + Carboplatin + Pemetrexed
Drug: Paclitaxel — Intravenous infusion
  Arms: Substudy B Phase 2 - Pumitamig Dose 1 + Carboplatin + Paclitaxel; Substudy B Phase 2 - Pumitamig Dose 2 + Carboplatin + Paclitaxel; Substudy B Phase 3 - Pembrolizumab + Carboplatin + Paclitaxel; Substudy B Phase 3 - Pumitamig + Carboplatin + Paclitaxel

SUMMARY:
This is a Phase 2/3, multisite, randomized, open-label study in participants with first-line non-small cell lung cancer (NSCLC).

This study includes two substudies (substudy A and substudy B) that will recruit participants according to histological subtypes due to differences in chemotherapy choice for standard-of-care and type of NSCLC.

DETAILED DESCRIPTION:
Each substudy contains a Phase 2 part followed by a Phase 3 part. Participants will be randomized to one of two dose levels of pumitamig (BNT327) plus chemotherapy for the Phase 2 part of each substudy. For the Phase 3 part of both substudies, an independent data monitoring committee (IDMC) and a blinded Independent Central Review (BICR) will be established. The IDMC will provide independent review of the data during the study as needed and the BICR will review all available tumor assessment scans for all treated participants.

The planned study duration per study participant is up to 64 months.

ELIGIBILITY:
Key Inclusion Criteria:

* Have systemic treatment naive, histologically or cytologically confirmed diagnosis of Stage IIIB or IIIC (who are not amenable to curative surgery or radiotherapy) or Stage IV NSCLC per the Union Internationale contre le Cancer/American Joint Committee on Cancer staging system, 9th edition.
* Have at least one measurable lesion as the targeted lesion based on RECIST v1.1. Lesions treated after prior local treatment (radiotherapy, ablation, interventional procedures, etc.) are generally not considered as target lesions. If the lesion with prior local treatment is the only targeted lesion, evidence-based radiology must be provided to demonstrate disease progression (the single bone metastasis or the single central nervous system metastasis should not be considered as a measurable lesion).
* Eastern Cooperative Oncology Group Performance Status of 0 or 1.
* Adequate organ function.

Key Exclusion Criteria:

* Have histologically or cytologically confirmed NSCLC with small-cell lung cancer histologic or neuroendocrine component.
* Have received any of the following therapies or drugs within the noted time intervals prior to study treatment:

  * Previous chemotherapy (platinum-based) or PD(L)-1 for treating NSCLC in either neo-adjuvant/adjuvant or locally advanced/metastatic setting.
  * Participants who received prior treatment with anti-VEGF monoclonal antibody, or PD(L)-1/VEGF bispecific antibody
  * Have received systemic corticosteroids (at a dosage greater than 10 mg/day of prednisone or an equivalent dose of other corticosteroids) within 7 days prior to the initiation of study treatment. Note: local, intranasal, intraocular, intra-articular or inhaled corticosteroids, short-term use (<=7 days) of corticosteroids for prophylaxis (e.g., prevention of contrast agent allergy) or treatment of non-autoimmune conditions (e.g., delayed hypersensitivity reactions caused by exposure to allergens) are allowed.
* Have uncontrolled hypertension or poorly controlled diabetic conditions prior to study treatment.
* Have a serious or non-healing wound, or (incompletely healed) bone fracture. This includes history (within 6 months prior to study entry) or risk of abdominal fistula, tracheoesophageal fistula, gastrointestinal perforation, or intra-abdominal abscess or esophageal and gastric varices. In addition, the participant must have undergone correction (or spontaneous healing) of the perforation/fistula and/or the underlying process causing fistula/perforation.
* Participants with significant risk of hemorrhage (per investigator clinical judgment).
* Have superior vena cava syndrome or symptoms of spinal cord compression.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1260 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Phase 2 - Occurrence of treatment-emergent adverse events (TEAE) (including Grade ≥3), adverse events of special interest (AESIs), treatment-related TEAEs, treatment-emergent serious adverse events (SAE), and treatment-related treatment emergent SAEs | From the first dose of the investigational medicinal product (IMP) to the 90-day Follow-Up Visit
  For substudies A and B. AEs graded according to Common Terminology Criteria for Adverse Events (CTCAE v5.0) in the combination treatment regimen.
Phase 2 - Occurrence of dose interruption, reduction, and discontinuation of IMP due to TEAEs (including related TEAEs) | From the first dose of IMP to the 90-day Follow-Up Visit
  For substudies A and B.
Phase 2 - Objective response rate (ORR) | Up to approximately 2 years
  For substudies A and B. ORR is defined as the proportion of participants in whom a confirmed complete response (CR) or confirmed partial response (PR) (per Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST v1.1] based on the investigator's assessment) is observed as best overall response.
Phase 2 - Best percentage change from baseline in tumor size | Up to approximately 2 years
  For substudies A and B. Based on investigator's tumor assessment according to RECIST v1.1.
Phase 3 - Progression free survival (PFS) assessed by blinded independent central review (BICR) | Up to approximately 5 years
  For substudies A and B. PFS defined as the time from randomization to first documented tumor progression (progressive disease per RECIST v1.1), or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Phase 3 - Overall survival (OS) | Up to approximately 5 years
  For substudies A and B. OS defined as the time from randomization to death from any cause
Phase 2 - Duration of Response (DOR) | Up to approximately 2 years
  For substudies A and B. DOR defined as the time from first objective response (CR or PR per RECIST v1.1) to first occurrence of objective tumor progression (progressive disease per RECIST v1.1) or death from any cause, whichever occurs first.
Phase 2 - Disease Control Rate (DCR) | Up to approximately 2 years
  For substudies A and B. DCR defined as the proportion of participants in whom a confirmed CR or confirmed PR or stable disease (per RECIST v1.1, stable disease assessed at least 6 weeks after randomization) is observed as best overall response.
Phase 3 - PFS assessed by investigator | Up to approximately 5 years
  For substudies A and B. PFS defined as the time from randomization to first documented tumor progression (progressive disease per RECIST v1.1), or death from any cause, whichever occurs first.
Phase 3 - ORR | Up to approximately 2 years
  For substudies A and B. ORR defined as the proportion of participants in whom a confirmed CR or confirmed PR (per RECIST v1.1) is observed as best overall response.
Phase 3 - PFS rate as assessed by BICR | At 6, 12, and 18 months
  For substudies A and B.
Phase 3 - PFS rate as assessed by investigator | At 6, 12, and 18 months
  For substudies A and B.
Phase 3 - OS rate | At 6, 12, 18, 24 months
  For substudies A and B.
Phase 3 - Change from baseline in European Organisation for Research and Treatment of Cancer (EORTC) Quality-of-life-score 30 Questionnaire (QLQ-C30) global health status/Quality-of-Life (QoL) score (Items 29 and 30) | Up to approximately 5 years
  For substudies A and B. The EORTC QLQ-C30 is the most widely used cancer-specific, health related QoL instrument containing a total of 30 items and measures 5 functional scales (physical, role, emotional, cognitive, and social), 3 symptom scales (fatigue, nausea/vomiting, and pain), 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties), and a global health status/QoL scale. All the scales and single-item measures range in score from 0 to 100 with a high scale score representing a higher response level (i.e., high score for global health status/QoL is high QoL: high score for symptom scale/item is high symptomatology or problems).
Phase 3 - Change from baseline in EORTC QLQ-C30 physical functioning | Up to approximately 5 years
  For substudies A and B. The EORTC QLQ-C30 is the most widely used cancer-specific, health related QoL instrument containing a total of 30 items and measures 5 functional scales (physical, role, emotional, cognitive, and social), 3 symptom scales (fatigue, nausea/vomiting, and pain), 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties), and a global health status/QoL scale. All the scales and single-item measures range in score from 0 to 100 with a high scale score representing a higher response level (i.e., high score for functional scale is high/healthy level of functioning).
Phase 3 - Change from baseline in coughing scale of the EORTC lung cancer-specific quality-of-life questionnaire (QLQ-LC29) | Up to approximately 5 years
  For substudies A and B. The EORTC QLQ-LC29 is a disease-specific supplementary health-related quality-of-life (HRQoL) questionnaire module to be employed in conjunction with the QLQ-C30. It comprises 29 items and measures five multi-item scales (coughing, shortness of breath, side effects, tumor progression/existential issues, surgery-related symptoms) and five single items (coughing up blood, pain in chest, arm/shoulder and other parts of the body, and weight loss). All the scales and single-item measures range in score from 0 to 100 with a high score for the scales and single items representing a high level of symptomatology or problems.
Phase 3 - Change from baseline in shortness of breath scale of the EORTC QLQ-LC29 | Up to approximately 5 years
  For substudies A and B. The EORTC QLQ-LC29 is a disease-specific supplementary health-related quality-of-life (HRQoL) questionnaire module to be employed in conjunction with the QLQ-C30. It comprises 29 items and measures five multi-item scales (coughing, shortness of breath, side effects, tumor progression/existential issues, surgery-related symptoms) and five single items (coughing up blood, pain in chest, arm/shoulder and other parts of the body, and weight loss). All the scales and single-item measures range in score from 0 to 100 with a high score for the scales and single items representing a high level of symptomatology or problems.
Phase 3 - Change from baseline in coughed up blood item of the EORTC QLQ-LC29 | Up to approximately 5 years
  For substudies A and B. The EORTC QLQ-LC29 is a disease-specific supplementary health-related quality-of-life (HRQoL) questionnaire module to be employed in conjunction with the QLQ-C30. It comprises 29 items and measures five multi-item scales (coughing, shortness of breath, side effects, tumor progression/existential issues, surgery-related symptoms) and five single items (coughing up blood, pain in chest, arm/shoulder and other parts of the body, and weight loss). All the scales and single-item measures range in score from 0 to 100 with a high score for the scales and single items representing a high level of symptomatology or problems.
Phase 3 - Change from baseline in fatigue domain score scale of the Non-Small Cell Lung Cancer Symptom Assessment Questionnaire (NSCLC-SAQ) | Up to approximately 5 years
  For substudies A and B. The NSCLC-SAQ is a 7-item patient-reported outcome measure for use in adults to assess symptoms of advanced non-small cell lung cancer. It contains five domains and accompanying items that were identified as symptoms of non small cell lung cancer: cough (1 item), pain (2), dyspnea (1), fatigue (2), and appetite (1). The (total) lowest score possible is 0, and the highest (total) score possible is 20. Higher scores indicate more severe symptoms.
Phase 3 - Change from baseline in pain domain score of the NSCLC-SAQ | Up to approximately 5 years
  For substudies A and B. The NSCLC-SAQ is a 7-item PRO measure for use in adults to assess symptoms of advanced non-small cell lung cancer. It contains five domains and accompanying items that were identified as symptoms of non small cell lung cancer: cough (1 item), pain (2), dyspnea (1), fatigue (2), and appetite (1). The (total) lowest score possible is 0, and the highest (total) score possible is 20. Higher scores indicate more severe symptoms.
Phase 3 - Change from baseline in Functional Assessment of Cancer Therapy-General item 5 overall bother item (FACT-GP5). | Up to approximately 5 years
  For substudies A and B. The FACT-G - Item GP5 (Version 4) is a single-item summary measure of the overall impact of treatment toxicity, based upon its association with the number and degree of AEs in clinical studies. The single-item GP5 ("I am bothered by side effects of treatment") is rated on a 5-point Likert scale ("not at all" to "very much") with a recall period of past 7 days.
Phase 3 - Occurrence of TEAEs including Grade ≥3, serious, and fatal TEAEs by relationship | From the first dose of IMP to the 90-day Follow-Up Visit
  For substudies A and B. AEs graded according to CTCAE v5.0.
Phase 3 - Occurrence of dose interruption, reduction, and discontinuation of IMP due to TEAEs (including related TEAEs) | From the first dose of IMP to the 90-day Follow-Up Visit
  For substudies A and B.

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (120):
- United States (19):
  - Alaska Oncology and Hematology, LLC, Anchorage, Alaska
  - Clermont Oncology Center, Clermont, Florida
  - H. Lee Moffit Cancer center and research institute, Tampa, Florida
  - Physicians Clinic of Iowa, Cedar Rapids, Iowa
  - Holden Comprehensive Cancer Center, University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Baptist Health Hardin, Elizabethtown, Kentucky
  - SSM Health Cancer Care - St. Clare, Fenton, Missouri
  - Mary Lanning Healthcare (MLH) - Morrison Cancer Center (MCC), Hastings, Nebraska
  - Astera Cancer Care, East Brunswick, New Jersey
  - The Valley Hospital - Valley Health System - The Robert and Audrey Luckow Pavilion, Paramus, New Jersey
  - White Plains Hospital, White Plains, New York
  - Fletcher Hospital, Inc. dba AdventHealth Hendersonville, Hendersonville, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - The Cleveland Clinic Cancer Center At Fairview Hospital, Moll Pavilion, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Cleveland Clinic - Hillcrest Hospital, Mayfield Heights, Ohio
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Baptist Cancer Center, Memphis, Tennessee
  - Millennium Research and Clinical Development, LLC, Houston, Texas
- Australia (10):
  - Cancer Research SA (CRSA), Adelaide
  - Royal Adelaide Hospital, Adelaide
  - Flinders Medical Centre, Bedford Park
  - Cairns Hospital, Cairns
  - Dubbo Hospital, Dubbo
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston
  - Icon Cancer Centre Kurralta Park, Kurralta Park
  - Western Health Sunshine Hospital, St Albans
  - ICON Cancer Care - Townsville, Townsville
  - Cancer Care Wollongong Pty Limited, Wollongong
- Belgium (2):
  - Universitair Ziekenhuis Leuven, Leuven
  - CHU HELORA, Hopital de Mons - Site Kennedy, Mons
- China (6):
  - Shandong University - Jinan Central Hospital, Jinan
  - Jiangsu Peoples Hospital, Nanjing
  - Shanghai Chest Hospital, Shanghai
  - Cancer Hospital of Shantou University Medical College, Shantou
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Chongqing University Three Gorges Hospital, Wanzhou
- France (7):
  - Centre Hospitalier Universitaire d'Angers (CHU Angers), Angers
  - Institut Bergonie - Centre Regional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux
  - CHU Caen Normandie, Caen
  - Centre Francois Baclesse, Caen
  - Centre Hospitalier Intercommunal de Creteil (CHIC) - Centre de ressources et de competences pour la mucoviscidose (C.R.C.M.), Créteil
  - Institut de Cancerologie de l'Ouest (ICO)- CRLCC Rene Gauducheau, Saint-Herblain
  - Centre Hospitalier Intercommunal Toulon La Seyne Sur Mer (C.H.I.T.S) - Hospital Font-Pre, Toulon
- Germany (6):
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - Asklepios Fachkliniken Muenchen Gauting, Gauting
  - Lungenfachklinik Immenhausen - Pneumologische Lehrklinik der Universitaet Goettingen, Immenhausen
  - MVZ for oncology and hematology Rhein-Kreis Neuss GmbH, Neuss
  - Praxiskooperation Bonn-Euskirchen-Rheinbach-Wesseling, Wesseling
  - Helios Klinikum Wuppertal-Universitaet Witten-Herdecke, Wuppertal
- Italy (9):
  - Azienda Ospedaliera San Giuseppe Moscati, Avellino
  - Centro di Riferimento Oncologico, Aviano
  - Ospedale San Luca, Lucca
  - IRCCS Istituto Romagnolo per lo studio dei Tumori Dino Amadori (IRST), Meldola
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale San Raffaele (HSR) (Istituto Scientifico Universitario San Raffaele), Milan
  - Casa Di Cura Polispecialistica Dott Pederzoli, Peschiera del Garda
  - Fondazione Policlinico Universitario Campus Bio-Medico, Roma
  - Fondazione Ospedale Isola Tiberina - Gemelli Isola, Rome
  - Universita di Siena -Azienda Ospedaliera Universitaria Senese-Policlincio Santa Maria Alle Scotte, Siena
- Tokyo Metropolitan Komagome Hospital, Bunkyō City, Japan
- Poland (3):
  - Instytut MSF Sp. z o.o., Lodz
  - NZOZ Medpolonia Sp. Z o.o., Poznan
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu, Przemyśl
- Romania (9):
  - Coltea Clinical Hospital, Bucharest
  - SC Gral Medical SRL, Bucharest
  - Cardiomed, Cluj-Napoca
  - S.C. Medisprof S.R.L, Oncologie medicala, Cluj-Napoca
  - Radiotherapy Center Cluj, Cluj-Napoca
  - Onco Clinic Consult SA, Craiova
  - Centrul de Oncologie Sf. Nectarie S.R.L (Sf Nectarie Oncology Center), Craiova
  - Ovidius Clinical Hospital, Ovidiu
  - Oncomed, Timișoara
- South Korea (11):
  - Chungbuk National University Hospital, Cheongju-si
  - Chungnam National University Hospital (CNUH), Daejeon
  - National Cancer Center, Goyang-si
  - Gachon University Gil Medical Center, Incheon
  - Gyeongsang National University Hospital (GNUH), Jinju
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center (AMC), Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - The Catholic University Of Korea, St. Vincent's Hospital, Suwon
  - Ajou University Hospital, Suwon
- Spain (6):
  - Consorcio Hospitalario Provincial de Castellón, Castellon
  - Complejo Hospitalario Universitario Insular Materno Infantil, Las Palmas de Gran Canaria
  - Hospital Universitari de Lleida Arnau de Villanova, Lleida
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Nuestra Senora De Valme, Seville
  - Hospital Universitario Miguel Servet de Zaragoza, Zaragoza
- Turkey (Türkiye) (22):
  - Adana City Training and Research Hospital, Adana
  - Gulhane Training and Research Hospital, Ankara
  - Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital, Ankara
  - Hacettepe University Medicine Faculty, Ankara
  - Memorial Ankara Hospital, Ankara
  - Liv Hospital Ankara, Ankara
  - Ankara Bilkent City Hospital, Ankara
  - Akdeniz University Hospital, Antalya
  - Gaziantep Sanko University Medical Faculty, Gaziantep
  - Bezmialem Foundation University Medical Faculty, Istanbul
  - Istinye University Bahcesehir Liv Hospital, Istanbul
  - Yeditepe University Kosuyolu Hospital, Istanbul
  - Medical Point Izmir Hospital, Izmir
  - Goztepe Prof. Dr. Suleyman Yalcin City Hospital, Kadıköy
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli
  - Medical Park Florya Hospital, Küçükçekmece
  - Sakarya University - Faculty of Medicine, Sakarya
  - Ondokuz Mayis University Health Practice and Research Hospital, Samsun
  - Acibadem Adana Hospital, Seyhan
  - Medical Park Seyhan Hospital, Seyhan
  - Gazi University Faculty of Medicine, Yenimahalle
  - Koc Universitesi Hastanesi (Koc University Hospital), Zeytinburnu
- United Kingdom (9):
  - Royal Sussex County Hospital - University Hospitals Sussex NHS Foundation Trust, Brighton
  - Velindre NHS Trust, Velindre Cancer Centre, Cardiff
  - Hull University Teaching Hospitals NHS Trust, Cottingham
  - University College Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Cancer And Haematology Centre-The Churchill Hospital-Oxford University Hospitals, Oxford
  - Royal Preston Hospital - Lancashire Teaching Hospitals NHS Foundation Trust, Preston
  - Southampton General Hospital, Southampton
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: No